CLINICAL TRIAL: NCT00681642
Title: Phase 1 Study of Comparison of the Effects on Promoting Corneal Epithelial Wound Healing Between Human Autoserum and Cord Blood Serum-in Vitro Cell Culture Experiment
Brief Title: Corneal Epithelial Wound Healing Difference Between Human Autoserum and Cord Blood Serum
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Wei-Li Chen, MD, PhD, Assistant Professor, National Taiwan University Hospital, department of Ophthalmology
Other Study IDs: 200702037R
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2010-12

CONDITIONS: Corneal Epithelial Wound Healing
Keywords: Corneal epithelial wound; Human autoserum; Cord blood

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Corneal epithelial tissue with wound cultured in human autoserum
- 2: Corneal epithelial tissue with wound cultured in umbilical cord serum

SUMMARY:
Human serum eye drops have been successfully used in the treatment of severe ocular surface disorders and the enhancement of corneal wound healing. Umbilical cord serum is also proven to be effective in treatment of dry eye and persistent corneal epithelial defects. However, there are limited studies comparing the corneal epithelial wound healing promoting effects between these two blood derived products. The purpose of this study is to test the corneal epithelial wound healing promoting effects between auto serum and human cord blood serum. Primary cultured bovine corneal epithelial cells were used as the model to investigate wound healing, cell proliferation and migration by means of scratch corneal wound healing assay evaluation, MTS assay and Boyden chamber migration assay in response to human serum and umbilical cord serum. The concentrations of EGF, TGF-β1, and fibronectin were also compared between human serum and umbilical cord serum with ELISA kits.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women
* Cesarean section for labor
* Complete placenta with umbilical cord retained
* Healthy individual

Exclusion Criteria:

* The retained placenta and umbilical cord were not complete
* Individual with anemia or other hematologic disorder unsuitable for blood donation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy pregnant women underwent smooth cesarean section during labor Healthy blood donor
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Cell proliferation | 1 week

SECONDARY OUTCOMES:
Cell migration | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Chen, MD, PhD, Principal Investigator — National Taiwan University Hospital, department of Ophthalmology
Locations (1):
- National Taiwan University Hospital, department of Ophthalmology, Taipei, Taiwan

REFERENCES:
- [Background] del Castillo JM, de la Casa JM, Sardina RC, Fernandez RM, Feijoo JG, Gomez AC, Rodero MM, Sanchez JG. Treatment of recurrent corneal erosions using autologous serum. Cornea. 2002 Nov;21(8):781-3. doi: 10.1097/00003226-200211000-00010. PMID 12410036
- [Background] Fox RI, Chan R, Michelson JB, Belmont JB, Michelson PE. Beneficial effect of artificial tears made with autologous serum in patients with keratoconjunctivitis sicca. Arthritis Rheum. 1984 Apr;27(4):459-61. doi: 10.1002/art.1780270415. No abstract available. PMID 6712760
- [Background] Geerling G, Maclennan S, Hartwig D. Autologous serum eye drops for ocular surface disorders. Br J Ophthalmol. 2004 Nov;88(11):1467-74. doi: 10.1136/bjo.2004.044347. PMID 15489495
- [Background] Goto E, Shimmura S, Shimazaki J, Tsubota K. Treatment of superior limbic keratoconjunctivitis by application of autologous serum. Cornea. 2001 Nov;20(8):807-10. doi: 10.1097/00003226-200111000-00006. PMID 11685056
- [Background] Poon AC, Geerling G, Dart JK, Fraenkel GE, Daniels JT. Autologous serum eyedrops for dry eyes and epithelial defects: clinical and in vitro toxicity studies. Br J Ophthalmol. 2001 Oct;85(10):1188-97. doi: 10.1136/bjo.85.10.1188. PMID 11567963
- [Background] Tsubota K, Goto E, Fujita H, Ono M, Inoue H, Saito I, Shimmura S. Treatment of dry eye by autologous serum application in Sjogren's syndrome. Br J Ophthalmol. 1999 Apr;83(4):390-5. doi: 10.1136/bjo.83.4.390. PMID 10434857
- [Background] Tsubota K, Goto E, Shimmura S, Shimazaki J. Treatment of persistent corneal epithelial defect by autologous serum application. Ophthalmology. 1999 Oct;106(10):1984-9. doi: 10.1016/S0161-6420(99)90412-8. PMID 10519596
- [Background] Tsubota K, Higuchi A. Serum application for the treatment of ocular surface disorders. Int Ophthalmol Clin. 2000 Fall;40(4):113-22. doi: 10.1097/00004397-200010000-00009. No abstract available. PMID 11064861
- [Background] Tsubota K, Satake Y, Ohyama M, Toda I, Takano Y, Ono M, Shinozaki N, Shimazaki J. Surgical reconstruction of the ocular surface in advanced ocular cicatricial pemphigoid and Stevens-Johnson syndrome. Am J Ophthalmol. 1996 Jul;122(1):38-52. doi: 10.1016/s0002-9394(14)71962-2. PMID 8659597
- [Background] Tsubota K, Shimazaki J. Surgical treatment of children blinded by Stevens-Johnson syndrome. Am J Ophthalmol. 1999 Nov;128(5):573-81. doi: 10.1016/s0002-9394(99)00224-x. PMID 10577524
- [Background] Yoon KC, Heo H, Jeong IY, Park YG. Therapeutic effect of umbilical cord serum eyedrops for persistent corneal epithelial defect. Korean J Ophthalmol. 2005 Sep;19(3):174-8. doi: 10.3341/kjo.2005.19.3.174. PMID 16209277
- [Background] Yoon KC, Im SK, Park YG, Jung YD, Yang SY, Choi J. Application of umbilical cord serum eyedrops for the treatment of dry eye syndrome. Cornea. 2006 Apr;25(3):268-72. doi: 10.1097/01.ico.0000183484.85636.b6. PMID 16633024
- [Background] Young AL, Cheng AC, Ng HK, Cheng LL, Leung GY, Lam DS. The use of autologous serum tears in persistent corneal epithelial defects. Eye (Lond). 2004 Jun;18(6):609-14. doi: 10.1038/sj.eye.6700721. PMID 15184926